CLINICAL TRIAL: NCT04186988
Title: Imaging of T-Cell Activation With [18F]-AraG in Advanced Non-Small Cell Lung Cancer (NSCLC) Patients Undergoing PD-1/PD-L1-Directed Therapy
Brief Title: [18F]-AraG for the Detection of T-Cell Activation in Advanced Non-small Cell Lung Cancer Patients Undergoing PD-1/PD-L1-Directed Therapy
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Unable to recruit to study.
Sponsor: University of California, Davis (Other)
Collaborators: National Cancer Institute (NCI) (NIH); CellSight Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1471901; NCI-2019-07768 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCHO030 (Other: University of California Davis Comprehensive Cancer Center); P30CA093373 (NIH)
Record Dates: First submitted 2019-12-02; First posted 2019-12-05 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Advanced Lung Non-Small Cell Carcinoma; Metastatic Lung Non-Small Cell Carcinoma; Stage III Lung Cancer AJCC v8; Stage IIIA Lung Cancer AJCC v8; Stage IIIB Lung Cancer AJCC v8; Stage IIIC Lung Cancer AJCC v8; Stage IV Lung Cancer AJCC v8; Stage IVA Lung Cancer AJCC v8; Stage IVB Lung Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Diagnostic ([18F]-AraG) (Experimental): Patients receive [18F]-AraG IV and then undergo PET/CT over 2 hours at baseline and within 2 weeks after starting immunotherapy. Patients may also undergo blood sample collection.
  Interventions: Drug: Fluorine F 18 Ara-G

INTERVENTIONS:
Drug: Fluorine F 18 Ara-G — Given IV
  Other Names: 18F-F-Ara-G; [18F]F-ara-G; [18F]F-AraG

SUMMARY:
This trial studies how well [18F]-AraG works in detecting T-cell activation in patients with non-small cell lung cancer that has spread to other places in the body (advanced), who are undergoing PD-1/PD-L1-directed therapy. [18F]-AraG is a "radiotracer" which attaches to immune cells directed at the cancer and shines a light that can be seen using a special camera, called a "positron emission tomography" or "PET" scanner. [18F]-AraG may improve the ability to detect a response of the cancer in the body to immunotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To quantify fluorine F 18 Ara-G ([18F]-AraG) uptake (standardized uptake value [SUV]) in advanced non-small cell lung cancer (NSCLC) tumor (primary, nodal, and metastatic sites) at baseline and after 1 dose of anti-PD-1/PD-L1 therapy in both patients treated with PD-1/PD-L1 monotherapy and in patients treated with immunotherapy/chemotherapy combination therapy.

II. To correlate change in [18F]-AraG uptake before and after the start of therapy with radiographic response in patients treated with immunotherapy.

OUTLINE:

Patients receive [18F]-AraG intravenously (IV) and then undergo PET/CT over 2 hours at baseline and within 2 weeks after starting immunotherapy. Patients may also undergo blood sample collection.

After completion of study treatment, patients are followed for up to 12 months.

ELIGIBILITY:
Inclusion Criteria:

* This study is open to all adult subjects with histological confirmation of NSCLC planned to undergo treatment with a PD-1 or PD-L1 inhibitor either as monotherapy or as combination therapy with concurrent chemotherapy as treatment for advanced/metastatic disease
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, 2 or 3 at the time of enrollment
* Patient with life expectancy >= 24 weeks from the time of screening to the study
* Ability to sign and understand the Institutional Review Board (IRB)-approved consent form in English
* Ability to remain motionless for up to 30 minutes per scan

Exclusion Criteria:

* Patients with severe claustrophobia (patients with milder forms of claustrophobia that can be successfully allayed with oral anxiolytic therapy are allowed)
* Severe impaired renal function with estimated glomerular filtration rate < 30 mL/min/1.73 m^2 and/or on dialysis
* Pregnancy
* Breast feeding an infant
* Prior treatment with anti-PD-1/PD-L1 inhibitor
* Localized/locally advanced disease with anti PD-1/PD-L1 given as consolidation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-11-05 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-03-12 (Actual)

PRIMARY OUTCOMES:
Fluorine F 18 Ara-G ([18F]-AraG) uptake values in advanced non-small cell lung cancer (NSCLC) before and after treatment with anti-PD-1/PD-L1 therapy obtained | Baseline up to within 2 weeks after starting immunotherapy
  The positron emission tomography (PET) images will be interpreted qualitatively and semi-quantitatively on a lesion-by-lesion basis. Semi-quantitative analysis will be employed as follows: (a) Regions of interest (ROIs) will be placed around tracer avid foci suspicious for malignancy in order to obtain standardized uptake value (SUV) parameters, including maximum SUV (SUVmax), SUVpeak, SUVmean; (b) SUV data will be recorded along with volumetric and positional information in a standardized form.

SECONDARY OUTCOMES:
Mean change in SUV | Baseline up to within 2 weeks after starting immunotherapy
  All SUV measurements will be summarized descriptively, separately for baseline and follow-up. Descriptive statistics for the SUVs will be done on a subject basis and a per lesion basis. Graphical summaries including box plots will be prepared to illustrate distributions and detect outliers or other findings; numerical summaries will include, mean, standard deviation (SD), median, and range as appropriate. For each target lesion, the scan 1 and scan 2 SUV will be determined and compared. A mixed-model repeated-measures analysis of variance (ANOVA) will be used to estimate the mean change in SUV from scan 1 to scan 2, allowing for possible need to account for between-patient random variation both in baseline level of SUV and amount of change. The primary result will be an estimate of the mean change in SUV, with a 95% confidence interval, along with the between patient and within-patient, between-lesion variation.
Correlation between [18F]-AraG uptake and clinical response | Baseline up to within 2 weeks after starting immunotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Julie Sutcliffe, Principal Investigator — University of California, Davis